CLINICAL TRIAL: NCT05958719
Title: Evaluation of Chidamide in Combination With Azacitidine, Liposomal Mitoxantrone, and Prednisone (CAMP Regimen) for Reviously Untreated Nodal T-follicular Helper (TFH) Cell Lymphoma
Brief Title: Chidamide in Combination With Azacitidine, Liposomal Mitoxantrone, and Prednisone (CAMP Regimen) for the Treatment of Previously Untreated Nodal TFH Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Zou Dehui, Assistant Director of lymphoma Diagnosis and Treatment Center, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023003
Record Dates: First submitted 2023-07-04; First posted 2023-07-25 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Peripheral T Cell Lymphoma; Epigenetic Repression
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Azacitidine; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interim evaluation of CR group (Experimental): Untreated patients with TFH-derived peripheral T-cell lymphoma will be treated with chidamide, azacitidine, liposomal mitoxantrone, and prednisone (CAMP regimen) for four cycles. For patients with interim-PET evaluation of CR, consolidation therapy with ASCT or another two cycles with CAMP regimen can be obtained. Subsequently,chidamide monotherapy was given as maintenance therapy for 24 months. Patients with interim evaluation of SD or PD withdrew from this study.
  Interventions: Drug: Chidamide; Drug: Azacitidine; Drug: liposomal mitoxantrone; Drug: prednisone
- interim evaluation of PR group (Experimental): Untreated patients with TFH-derived peripheral T-cell lymphoma will be treated withchidamide, azacitidine, liposomal mitoxantrone, and prednisone (CAMP regimen) for four cycles. For patients with interim-PET evaluation of PR, another two cycles of CAMP regimen will be continued, followed by the second PET-CT efficacy evaluation, and those who achieve CR receive consolidation therapy with ASCT and following chidamide maintenance. Subsequently, chidamide monotherapy was given as maintenance therapy for 24 months. Patients with second efficacy evaluation of PR or SD or PD withdrew from this study.
  Interventions: Drug: Chidamide; Drug: Azacitidine; Drug: liposomal mitoxantrone; Drug: prednisone

INTERVENTIONS:
Drug: Chidamide — chidamide 30mg biw, p.o, 21 days for a cycle.
Drug: Azacitidine — 75mg/m2, continuous i.h. on day 1-7，21 days for a cycle.
Drug: liposomal mitoxantrone — 12mg/m2， d1,21 days for a cycle.
Drug: prednisone — 60mg/m2，d1-5,21 days for a cycle.

SUMMARY:
This study is investigating the effectiveness (specifically the objective response rate - ORR) of a new combination therapy called CAMP (chidamide, azacitidine, liposomal mitoxantrone, and prednisone) for previously untreated angioimmunoblastic T-cell lymphoma (AITL). It's a single-arm study comparing CAMP's safety and efficacy to standard treatments. Younger patients (≤70) receive the full CAMP regimen, while older patients receive a modified version (CAMP-light). Patients are assessed via PET-CT after 4 cycles. Responders (CR/PR) receive consolidation therapy and then maintenance chidamide for 2 years. Eligible patients achieving CR after 4 cycles can get a transplant, while those with PR need 2 more cycles first. Patients with stable or progressive disease after 4 cycles are withdrawn. Progression at any time leads to study discontinuation.

DETAILED DESCRIPTION:
Main Objective:

The primary objective of this study is to investigate the objective response rate (ORR) of chidamide in combination with azacitidine, liposomal mitoxantrone, and prednisone (CAMP regimen) for the treatment of treatment-naïve angioimmunoblastic T-cell lymphoma (AITL).

Study Design:

This study employs a single-arm design, based on the hypothesis that the safety profile of the chidamide, azacitidine, liposomal mitoxantrone, and prednisone (CAMP regimen) is superior to conventional treatment regimens, and that the efficacy, as measured by ORR, is non-inferior to conventional treatment regimens. Patients meeting the inclusion/exclusion criteria will be treated according to age: patients ≤70 years old will receive the CAMP regimen as first-line therapy, while patients >70 years old will receive a modified CAMP regimen (CAMP-light) as first-line therapy. Interim efficacy will be assessed via PET-CT scan after the 4th cycle of chemotherapy, with PET-CT results interpreted using the Deauville 5-point scale.

Treatment and Follow-up:

Patients achieving a complete response (CR) or partial response (PR) at the interim assessment will continue with 2 cycles of consolidation therapy using the CAMP regimen or CAMP-light regimen. Subsequently, they will enter single-agent chidamide maintenance therapy (≤70 years old: chidamide 30mg orally, twice weekly; >70 years old: chidamide 20mg orally, twice weekly), which will continue for 24 months.

Patients eligible for transplantation who achieve a CR after 4 cycles of induction therapy may proceed to autologous stem cell transplantation (ASCT). Patients achieving a PR will receive 2 additional cycles of consolidation therapy before undergoing ASCT. Patients with a PR at the interim assessment will undergo a repeat PET-CT scan before transplantation to reassess efficacy. Stem cell mobilization for transplant-eligible patients will utilize steady-state mobilization with or without plerixafor.

Patients exhibiting stable disease (SD) or progressive disease (PD) at the interim assessment after 4 cycles will be withdrawn from the study.

Patients experiencing PD at any time during the treatment course will be discontinued from the study upon confirmation of progression.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histological confirmation of nodal T-follicular helper (TFH) cell lymphoma.
2. More than 18 years of age.
3. Proper functioning of the major organs: 1) The absolute value of neutrophils (≥1×10^9/L); 2) platelet count (≥75×10^9/L); 3) Serum total bilirubin ≤ 1.5 times ULN; 4) Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) ≤3 times ULN; 5) Serum creatinine (Cr) ≤2 ULN, or glomerular filtration rate ≥40ml/min;
4. Eastern Cooperative Oncology Group (ECOG) Performance status 0-2.
5. LVEF value measured by echocardiography ≥50%.
6. Life expectancy > 3 months.

Exclusion Criteria:

1. Patients who have previously received chemotherapy, radiotherapy or other antitumor therapy.
2. Patients with central nervous system involvement by lymphoma.
3. Patients with uncontrolled cardiovascular and cerebrovascular diseases, coagulation disorders, connective tissue diseases, serious infectious diseases and other diseases.
4. Pregnant or breastfeeding women.
5. Presence of human immunodeficiency virus (HIV) virus infection.
6. Previous history of other malignant tumors, unless the disease has been cured for 5 years or more. The following cured tumors are excluded:

   1. Basal cell carcinoma of the skin, squamous cell carcinoma of the skin and related localized non-melanoma skin cancers;
   2. Carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years post initiation of treatment
  ORR is defined as the incidence of either a CR or a partial response (PR) per the Lugano Classification by PET-CT as determined by study investigators.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 2 years post initiation of treatment

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years post initiation of treatment
  PFS is defined as the time from the initiation of treatment to the date of disease progression or death from any cause.
Duration of Response (DOR) | 2 years post initiation of treatment
  DOR is defined for participants who experience complete response after treatment and is the time from the first objective response to disease progression or death from any cause.
Overall Survival (OS) | 2 years post initiation of treatment
  OS is defined as the time from initiation of treatment to the date of death from any cause.

OTHER OUTCOMES:
levels of lymphocyte subsets in blood | 2 years post initiation of treatment
levels of cytokines in serum | 2 years post initiation of treatment
  Cytokines assessed by flow cytometry: including IL-10, IL-6, IL-8, IFN-α, IFN-γ, and TNF-α.

CONTACTS AND LOCATIONS:
Overall Officials: Dehui Zou, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No